CLINICAL TRIAL: NCT01591005
Title: Risk Reduction of Symptomatic and Silent Brain Infarctions During Carotid Endarterectomy and Carotid Stenting Due to Ultrasound Activation of Endogenous Fibrinolytic System Using Transcranial Doppler Monitoring
Brief Title: SONOlysis in Prevention of Brain Infarctions dUring Carotid Stenting and caroTid EndaRterectomy
Acronym: SONOBUSTER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: Palacky University (Other)
Responsible Party: Principal Investigator, Vaclav Prochazka, MD, PhD. MSc, Vaclav Prochazka, MD, PhD, MSc, University Hospital Ostrava
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NT11386-5/2010
Record Dates: First submitted 2012-04-23; First posted 2012-05-03 (Estimated); Results first posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-07

CONDITIONS: Internal Carotid Artery Stenosis
Keywords: sonolysis; carotid; endarterectomy; stenting
MeSH Terms: conditions — Carotid Stenosis | interventions — Endarterectomy; Endarterectomy, Carotid; Angioplasty; Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CEA with sonolysis (Experimental): endarterectomy with sonolysis (continual transcranial Doppler monitoring)
  Interventions: Procedure: sonolysis; Procedure: endarterectomy
- CEA without sonolysis (Placebo Comparator): endarterectomy without sonolysis
  Interventions: Procedure: endarterectomy
- carotid stenting with sonolysis (Experimental): carotid stenting with sonolysis (continual transcranial Doppler monitoring)
  Interventions: Procedure: sonolysis; Procedure: carotid stenting
- carotid stenting without sonolysis (Placebo Comparator): carotid stenting without sonolysis
  Interventions: Procedure: carotid stenting

INTERVENTIONS:
Procedure: sonolysis — continual transcranial Doppler monitoring with max. diagnostic intensity for 60 minutes
  Other Names: sonothrombolysis; sonothrombotripsy
  Arms: CEA with sonolysis; carotid stenting with sonolysis
Procedure: endarterectomy — carotid endarterectomy
  Other Names: carotid endarterectomy
  Arms: CEA with sonolysis; CEA without sonolysis
Procedure: carotid stenting — percutaneous transluminal angioplasty and stenting
  Other Names: percutaneous transluminal angioplasty and stenting
  Arms: carotid stenting with sonolysis; carotid stenting without sonolysis

SUMMARY:
The aim of the project is to demonstrate a fibrinolytic effect of sonothrombolysis (continual transcranial Doppler monitoring) using 2 MegaHertz (MHz) diagnostic probe on the reduction of risk of brain infarctions due to the activation of endogenous fibrinolytic system during carotid endarterectomy (CEA) and carotid stenting (CS). 240 patients indicated for CEA (120 patients) and CS (120 patients) will be enrolled into the study in order to demonstrate a twenty-percent risk reduction of number and volume of brain infarctions detected using MRI examination 24 hours after CEA or CS in 5% level of significance. Patients will be randomized - subgroup 1 will undergo a 60minute non-diagnostic transcranial Doppler (TCD) monitoring during CEA or CS, subgroup 2 will undergo interventions without TCD monitoring. The second aim is to compare number of brain infarctions detected using MRI between CEA and CS patients.

Confirmation of the investigators hypothesis that sonothrombolysis is able to activate endogenous fibrinolytic system during CEA or CS with consecutive reduction of the number and volume of brain infarcts, can lead to the increase of the safety of CEA and CS in patients with internal carotid artery stenosis. The investigators can presume that up to 50% of patients indicated for CEA or CS can be treated using these methods in the future.

In the Substudy "Risk of brain infarction after carotid endarterectomy and stenting" the the risk of asymptomatic and symptomatic brain infarctions, changes in cognitive functions, as well as morbidity and mortality at 30 days between patients with symptomatic and asymptomatic severe internal carotid artery (ICA) stenoses undergoing elective CEA and CAS will be compared.

The sample size of the Substudy was based on an expected 80% difference of new ischemic lesions on DWI-MRI between CEA (estimated prevalence, 30%) and CAS (54%). Pre-study calculations showed that a minimum of 73 patients in each group was needed to reach a significant difference with an alpha value of 0.05 (two-tailed) and a beta value of 0.8 assuming that 15% of subjects would be lost to follow-up or refuse to participate in the study.

DETAILED DESCRIPTION:
AIM OF THE PROJECT AND HYPOTHESIS The aim of the project is to demonstrate an effect of continual TCD monitoring using 2 MHz diagnostic probe with maximal diagnostic energy on the reduction of risk of brain microinfarctions due to the activation of endogenous fibrinolytic system during CEA and CS. The second aim of the study is to compare the risk of brain infarction between CEA and CS.

240 patients indicated for CEA (120 patients) and CS (120 patients) will be enrolled into the study in order to demonstrate a twenty-percent risk reduction of number and volume of brain infarctions detected using MRI examination 24 hours after CEA or CS in 5% level of statistical significance. Patients will be randomized into 2 subgroups. Subgroup 1 will undergo a 60minute non-diagnostic TCD monitoring during CEA or CS. Subgroup 2 will undergo CEA or CS without TCD monitoring. The second aim is to compare number and volume of brain infarctions detected using MRI between CEA and CS patients.

Substudy "Risk of brain infarction after carotid endarterectomy and stenting" The aim of the prospective, randomized study was to compare the risk of asymptomatic and symptomatic brain infarctions, changes in cognitive functions, as well as morbidity and mortality at 30 days between patients with symptomatic and asymptomatic severe ICA stenoses undergoing elective CEA and CS.

PATIENTS AND METHODS 240 patients with ICA stenosis indicated for CEA or CS according to the criteria of the American Heart Association will be enrolled into the study during a 4-year period. Altogether 120 patients indicated for CEA and 120 patients indicated for CS will be randomized for standard CEA / CS and TCD monitored CEA / CS.

Randomization: Randomization using computer generated random allocation will be used, separately for CEA and CS patients.

Substudy "Risk of brain infarction after carotid endarterectomy and stenting" Minimally146 patients with ICA stenosis >70% (symptomatic or asymptomatic) detected by duplex sonography and confirmed using computed tomography angiography (CTA); indication for carotid intervention (CEA or CAS) according to criteria set by the American Heart Association5; age 40-80 years; (iv) functionally independent (modified Rankin score 0-2 points); no contraindication to magnetic resonance imaging (MRI), computer tomography angiography (CTA) or digital angiography (DSA) will be enrolled to the Substudy.

Randomization: Randomization using computer generated random allocation to CEA or CS will be used.

Sonothrombolysis: In patients randomized into sonothrombolysis subgroup, middle cerebral artery (MCA) segment in depth 55 mm will be monitored for 40 minutes using a diagnostic 2 MHz probe with maximal diagnostic energy. Non-diagnostic TCD monitoring will be performed without detection of microembolic signals or detection of changes in blood flow. The second (control) subgroup will undergo a standard CEA or CS without sonothrombolysis.

MRI protocol will consists of 4 sequences: 1. Localizer; 2. T2-weighted images (T2TSE); 3. fluid-attenuated inversion recovery (FLAIR); 4. diffusion-weighted imaging (DWI). Sequences 1-3 will be applied in the same level, they will have the same slice thickness and the same cut number. The slice thickness comprises its own cut thickness (5 mm) + distant factor (30%). Standard number of slices is 19. Standard slice level is considered to be a modified level of skull base due to the minimalization of distant artifacts echo planar imaging (EPI) sequence. Sequence called "trace" with three types of magnetic resonance pictures in every slice: (a) T2*EPI b=0; (b) DWI b=500; (c) DWI b=1000. The fourth type of images automatically created an apparent diffusion coefficient (ADC) map (in-line postprocessing). DWI show a middle (average) diffusivity of every point of examined brain tissue when b value is 500 and 1000. This sequence is applied in order to assess hemorrhage (T2*EPI) and monitor sites of reduced diffusion (DWI, b=500 and 1000). New infarctions will be evaluated only in the territory of treated ICA.

Adverse effects: All adverse effects during 1 month after ultrasound monitoring will be registered, especially all causes for new admissions to the hospital, worsening of neurological symptoms (>4 points in NIH stroke scale), brain edema, symptomatic and asymptomatic intracranial bleeding detected in control brain MRI.

Statistic evaluation: All statistical tests will be performed at the Department of Biophysics, Informatics and Biometry, Palacký University Medical School, Olomouc. Statistical evaluation in 5% level of significance of differences in the number and volume of brain infarctions detected using MRI between patients with TCD monitoring and without TCD monitoring during CEA or CS will be performed using Student T-test, χ2-test, Mann-Whitney U-test, ANOVA and multivariate analysis. Differences in the number and volume of brain infarctions between patients after CEA and CS will be evaluated as secondary end-points. Influence of other factors, e.g. age, gender, symptoms in the territory of treated artery, number of infarctions before CEA or CS, results of cognitive tests will be evaluated.

Statistic evaluation for Substudy: The normality of distribution of all data will be checked using the Shapiro-Wilk test. Categorical variables in the two arms will be compared by Fisher's exact test. Continuous variables will be compared by the Student's t-test for normally distributed values and by Mann-Whitney U test for other values. Multiple logistic regression analyses were used to determine the possible predictors of a new brain infarction. All tests were carried out at an alpha level of significance of 0.05.

Study protocol has been approved by the Ethics Committees in accordance with the principles and guidelines of the Declaration of Helsinki, 1975.

ELIGIBILITY:
Inclusion Criteria:

* stenosis of internal carotid artery
* indication to endarterectomy or stenting
* age 40-80 years
* sufficient temporal bone window for TCD with detectable blood flow in MCA
* independent patient (modified Rankin score 0-2)
* informed consent signed by the patient.

Exclusion Criteria:

* contraindication to MRI examination (pace-maker, implanted metal material, claustrophobia)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2010-10; Primary Completion 2014-07 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Skoloudik, MD, PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Skoloudik D, Kuliha M, Hrbac T, Jonszta T, Herzig R; SONOBUSTER Trial Group. Sonolysis in Prevention of Brain Infarction During Carotid Endarterectomy and Stenting (SONOBUSTER): a randomized, controlled trial. Eur Heart J. 2016 Oct 21;37(40):3096-3102. doi: 10.1093/eurheartj/ehv492. Epub 2015 Sep 28. PMID 26417059
- [Derived] Kuliha M, Roubec M, Prochazka V, Jonszta T, Hrbac T, Havelka J, Goldirova A, Langova K, Herzig R, Skoloudik D. Randomized clinical trial comparing neurological outcomes after carotid endarterectomy or stenting. Br J Surg. 2015 Feb;102(3):194-201. doi: 10.1002/bjs.9677. Epub 2014 Dec 16. PMID 25511816
- See also: University Hospital Ostrava — http://fno.cz
- See also: Ministry of Health of Czech Republic — http://mzcr.cz

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CEA With Sonolysis | CEA Without Sonolysis | Carotid Stenting With Sonolysis | Carotid Stenting Without Sonolysis
Started | 53 | 53 | 68 | 68
Completed | 53 | 53 | 68 | 68
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: In total, 242 of the 495 screened patients fulfilled the inclusion criteria. Subjects were randomly and equally allocated to the sonolysis or control group. Clinical and procedural variables were well balanced between the groups
Groups:
- Total: Total of all reporting groups
Arm/Group | CEA With Sonolysis | CEA Without Sonolysis | Carotid Stenting With Sonolysis | Carotid Stenting Without Sonolysis | Total
Number analyzed (Participants) | 53 | 53 | 68 | 68 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (7.3) | 63.0 (7.5) | 66.8 (6.7) | 68.5 (7.7) | 65.8 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 15 | 24 | 80
  Male | 33 | 32 | 53 | 44 | 162
Region of Enrollment [Number; unit: participants]
  Czech Republic | 53 | 53 | 68 | 68 | 242

OUTCOME MEASURES:

1. Primary Outcome: Participants With a New Brain Infarction Detected Using Magnetic Resonance
Description: The number of participants with a new brain infarctions in sonolysis group detected using magnetic resonance examination 24 hours after carotid endarterectomy or carotid stenting.
  Substudy: The number of participants with a new brain infarctions on brain diffusion-weighted magnetic resonance imaging performed 24 hours after intervention in carotid endarterectomy and carotid stenting groups.
Time Frame: 24 hours after intervention
Measure: Number; unit: participants
Groups:
- Carotid Endarterectomy With Sonolysis: endarterectomy with sonolysis (continual transcranial Doppler monitoring)
  sonolysis: continual transcranial Doppler monitoring with max. diagnostic intensity for 60 minutes
  endarterectomy: carotid endarterectomy
- Carotid Endarterectomy Without Sonolysis: endarterectomy without sonolysis
  endarterectomy: carotid endarterectomy
Arm/Group | Carotid Endarterectomy With Sonolysis | Carotid Endarterectomy Without Sonolysis | Carotid Stenting With Sonolysis | Carotid Stenting Without Sonolysis
Number analyzed (Participants) | 53 | 53 | 68 | 68
participants | 5 | 15 | 33 | 42

2. Secondary Outcome: Participants With a New Brain Infarctions Detected Using Magnetic Resonance in Endarterectomy and Stenting Groups
Description: The number of participants with a new brain infarctions >0.5 cm3 detected using magnetic resonance examination 24 hours after intervention between endarterectomy and stenting using periprocedural sonolysis.
  Substudy: The number of participants with a new brain infarctions >0.5 cm3 detected using magnetic resonance examination 24 hours after intervention between carotid endarterectomy and carotid stenting groups.
Time Frame: 24 hours after intervention
Measure: Number; unit: participants
Arm/Group | Carotid Endarterectomy With Sonolysis | Carotid Endarterectomy Without Sonolysis | Carotid Stenting With Sonolysis | Carotid Stenting Without Sonolysis
Number analyzed (Participants) | 53 | 53 | 68 | 68
participants | 3 | 7 | 3 | 17

3. Secondary Outcome: Cognitive Decline
Description: The changes in cognitive functions after carotid endarterectomy and carotid stenting measured by Mini-Mental State Examination using periprocedural sonolysis.
  Substudy: The changes in cognitive functions after intervention measured by Mini-Mental State Examination between carotid endarterectomy and carotid stenting groups.
  Range of scores possible for the Mini-Mental State Examination: 0 - 30 points. Higher values in this range are considered to be a better outcome.
Time Frame: 24 hours after intervention
Population: only patients with performed Mini Mental State examination
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Carotid Endarterectomy With Sonolysis | Carotid Endarterectomy Without Sonolysis | Carotid Stenting With Sonolysis | Carotid Stenting Without Sonolysis
Number analyzed (Participants) | 35 | 37 | 47 | 46
Scores on a scale | 28 [26 to 29] | 27 [25 to 28] | 28 [26 to 29] | 27 [25 to 29]

4. Secondary Outcome: Number of Participants With Clinical Manifested Brain Infarction
Description: The risk of stroke or transient ischemic attack (at 24 hours and 30 days) due to the activation of endogenous fibrinolytic system during carotid endarterectomy and carotid stenting using periprocedural sonolysis.
  Substudy: The risk of stroke or transient ischemic attack (at 24 hours and 30 days) due to the activation of endogenous fibrinolytic system between carotid endarterectomy and carotid stenting groups.
Time Frame: 24 hours and 30 days after intervention
Measure: Number; unit: participants
Arm/Group | Carotid Endarterectomy With Sonolysis | Carotid Endarterectomy Without Sonolysis | Carotid Stenting With Sonolysis | Carotid Stenting Without Sonolysis
Number analyzed (Participants) | 53 | 53 | 68 | 68
participants | 1 | 0 | 0 | 3

5. Secondary Outcome: Number of Participatns With New Ipsilateral Brain Infarctions Detected Using MRI in Endarterectomy and Stenting Groups
Description: The number of patients with the ipsilateral brain infarctions detected using MRI examination 24 hours after intervention between endarterectomy and stenting using periprocedural sonolysis.
  Substudy: The number of patients with the ipsilateral brain infarctions detected using MRI examination 24 hours after intervention between carotid endarterectomy and carotid stenting groups.
Time Frame: 24 hours after intervention
Measure: Number; unit: participants
Arm/Group | Carotid Endarterectomy With Sonolysis | Carotid Endarterectomy Without Sonolysis | Carotid Stenting With Sonolysis | Carotid Stenting Without Sonolysis
Number analyzed (Participants) | 53 | 53 | 68 | 68
participants | 5 | 14 | 26 | 38

6. Secondary Outcome: Number of Participants With Clinical Vascular Event or Death
Description: The risk of the occurrence of death, any stroke, or myocardial infarction within 30 days (myocardial infarction was defined as a post-interventional cardiac troponin T level increase >2-fold the upper limit of normal in addition to either chest pain or symptoms consistent with ischemia or electrocardiographic evidence of ischemia) after carotid endarterectomy and carotid stenting using periprocedural sonolysis.
  Substudy: The risk of the occurrence of death, any stroke, or myocardial infarction within 30 days (myocardial infarction was defined as a post-interventional cardiac troponin T level increase >2-fold the upper limit of normal in addition to either chest pain or symptoms consistent with ischemia or electrocardiographic evidence of ischemia) between carotid endarterectomy and carotid stenting groups.
Time Frame: 30 days after intervention
Measure: Number; unit: participants
Arm/Group | Carotid Endarterectomy With Sonolysis | Carotid Endarterectomy Without Sonolysis | Carotid Stenting With Sonolysis | Carotid Stenting Without Sonolysis
Number analyzed (Participants) | 53 | 53 | 68 | 68
participants | 0 | 0 | 0 | 0

7. Other Pre Specified Outcome: Number of Participants With Complications
Description: Any complication during carotid endarterectomy and carotid stenting, sonolysis or 30 days after intervention in all subgroups.
Time Frame: 24 hours and 30 days after intervention
Measure: Number; unit: participants
Arm/Group | Carotid Endarterectomy With Sonolysis | Carotid Endarterectomy Without Sonolysis | Carotid Stenting With Sonolysis | Carotid Stenting Without Sonolysis
Number analyzed (Participants) | 53 | 53 | 68 | 68
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | CEA With Sonolysis | CEA Without Sonolysis | Carotid Stenting With Sonolysis | Carotid Stenting Without Sonolysis
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/68 | 0/68

LIMITATIONS AND CAVEATS:
Serial follow-up MRI was not done. A software package for mapping of brain infarction volume was not used. Single-centre investigation with mandatory use of brain protection device during carotid stenting and shunt during carotid endarterectomy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes